CLINICAL TRIAL: NCT04763590
Title: Cognitive Behavioral Therapy for Mechanical Ventilation Wean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 828187
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Anxiety; Cognitive Behavioral Therapy; Mechanical Ventilation Complication
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy (Experimental): Cognitive Behavioral Therapy (CBT) had 3 principal components: (1) psychoeducation, (2) cognitive restructuring, and (3) exposure. In this treatment, derived from an empirically-supported treatment for panic disorder, psychoeducation consisted of teaching about the interrelationship between thoughts, feelings, and physical sensations during weaning. The cognitive component taught patients how to challenge their thoughts, with a particular focus on identifying thoughts that over-estimated the probability of negative medical events. The behavioral component consisted of reducing the need for mechanical ventilation in a step-wise, graduated, manner.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — This study focuses on patients who are on a mechanical ventilator and who have been medically cleared to come off of it. The purpose of the study is to learn more about the possible influence of cognitive behavioral therapy in helping patients who are having some trouble getting off of the ventilator. Cognitive behavioral therapy is a highly effective intervention for anxiety and the investigators are evaluating whether cognitive behavioral therapy might be helpful in cases where it is difficult to come off of the ventilator.
  Cognitive behavioral therapy is experimental for mechanical ventilation assistance as no research to date has evaluated whether it might be helpful.

SUMMARY:
The purpose of this study is to use CBT strategies in assisting patients hospitalized in intensive care units in ventilation wean through a case series of 2 patients.

DETAILED DESCRIPTION:
Approximately a third of patients in intensive care are mechanically ventilated. The current weaning standard of care leaves much to be desired in both patient anxiety and time to wean. Cognitive behavioral therapy (CBT) is the gold standard treatment for anxiety. The purpose of this study is to use CBT strategies in assisting patients hospitalized in intensive care units in ventilation wean through a case series of 2 patients.

ELIGIBILITY:
Inclusion Criteria:

* Receiving mechanical ventilation and Failed 3 spontaneous breathing trials

Exclusion Criteria:

* Delirium

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Respiratory Anxiety | 6 weeks
  The Anxiety Inventory for Respiratory Disease provides an assessment of anxiety in patient with respiratory disease which is free of the physical symptoms of respiratory disease that often overlap with and confound an accurate assessment of anxiety. A score of 14.5 discriminates between patients with and without anxiety. The measure is reliable, valid, and sensitive to change.
Panic Symptoms | 6 weeks
  the investigators assessed whether patients experienced the panic symptoms listed in the Diagnostic and Statistical Manual of Mental Disorders, 5th edition, when weaning from the ventilator or when anticipating weaning and, if they endorsed the symptom, asked patients to rate symptom severity from 1 to 7 (7 being the worst).
Generalized Anxiety | 6 weeks
  The investigators assessed generalized anxiety with the Generalized Anxiety Disorder 7 Scale (GAD-7). The minimum score is zero and maximum score is 21. Higher scores represent a worse outcome. A score of 10 on the Generalized Anxiety Disorder 7 represents clinically significant levels of generalized anxiety.
Depression | 6 weeks
  The investigators assessed depression with the Patient Health Questionnaire 2 (PHQ-2). The scale ranges from zero to 6, with higher scores representing a worse outcome. A score of 3 or higher signifies likely clinical depression.
Time spent on tracheostomy-collar (off mechanical ventilation) | 6 weeks
  Time on tracheostomy collar (TC) was assessed from the beginning of the cognitive behavioral therapy intervention until study completion.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen JN, Gopal A, Roberts KJ, Anderson E, Siegel AM. Ventilator-Dependent Patients Successfully Weaned With Cognitive-Behavioral Therapy: A Case Series. Psychosomatics. 2019 Nov-Dec;60(6):612-619. doi: 10.1016/j.psym.2019.02.003. Epub 2019 Feb 12. No abstract available. PMID 31327505